CLINICAL TRIAL: NCT05970484
Title: Supporting Women in the UK Armed Forces Who Consume Alcohol at an Increased Risk: Refining the DrinksRation Platform - Study Protocol
Brief Title: Supporting Women in the UK Armed Forces Who Consume Alcohol at an Increased Risk: Refining the DrinksRation Platform
Acronym: RationW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Lancaster University (Other); Combat Stress (Other); Swansea University (Other); UK British Army (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: LRS/DP-22/23-36879
Record Dates: First submitted 2023-07-24; First posted 2023-08-01 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Abuse; Alcohol Drinking; Alcohol Use Disorder
Keywords: digital health
MeSH Terms: conditions — Alcoholism; Alcohol Drinking

STUDY DESIGN:
Intervention Model Description: This is a two-arm participant-blinded (single-blinded) confirmatory randomized controlled trial (RCT), comparing (intervention arm) the DrinksRation smartphone app with (control arm) a progressive web application (PWA) presenting NHS-focused drinking advice (named 'BeAlcoholSmart'). The DrinksRation app provides individualized normative advice with features designed to enhance participant motivation, interactive feedback, self-efficacy in modifying their alcohol consumption, and personalized gender-specific messaging. We hypothesize that the intervention arm will be efficacious in reducing alcohol consumption compared with the control arm.
Who Masked: Participant, Investigator
Masking Description: Researcher DL and GW will be unblinded to treatment allocation to enable the management of the BeAlcoholSmart and DrinksRation platforms and participant recruitment and retention; researcher EC will be unblinded to treatment allocation to prepare statistical reports. Researcher DL and EC will not be involved in participant engagement. All other members of the study team will be blind to treatment allocation.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Use of the DrinksRation app with all functionality
  Interventions: Behavioral: DrinksRation
- Control (Active Comparator): Use of the BeAlcoholSmart app with all functionality
  Interventions: Behavioral: BeAlcoholSmart

INTERVENTIONS:
Behavioral: DrinksRation — DrinksRation (www.drinksration.app; formerly called InDEx) app was developed following the Medical Research Council Complex Intervention Guidelines and using a co-design methodology. It was developed by the King's Centre for Military Health Research (King's College London) and Lancaster University, supported by experts in smartphone app development, epidemiology, addiction psychiatry, and military mental health. The app was designed to support veterans drinking at a hazardous or harmful level by providing bespoke advice and support.
  Arms: Intervention
Behavioral: BeAlcoholSmart — BeAlcoholSmart is a progressive web app (PWA). The app can take advantage of smartphone features such as push notifications and haptics without requiring the participant to download via an app store. The app will contain a 7-day alcohol unit calculator and generic public health guidance on safe drinking. Participants will also receive reminders via email prompting them to consult the guidance as part of the BeAlcoholSmart. Control participant participants will be invited to complete all questionnaires via Qualtrics, with an email reminder being sent when they are due.
  Arms: Control

SUMMARY:
Alcohol misuse is common in the Armed Forces (AF), with prevalence higher than in the general population. To date, initiatives to support alcohol misuse have focused on males, who represent ~90% of the AF. However, female veterans drink disproportionally more than female members of the public. In this study, the investigators will refine and evaluate DrinksRation - the only automated brief digital intervention supporting the United Kingdom (UK) Armed Forces to manage and reduce the amount they drink - to tailor the intervention to the specific needs of female veterans. The changes will then be assessed using a confirmatory Randomized Controlled Trial (RCT), which includes a minimum of 148 (74 in each arm) female veterans (to be recruited).

DETAILED DESCRIPTION:
There are 2.5 million AF veterans in the UK (defined by the British Government as those who have served in the military for at least one paid day), of which 11% are estimated to identify as female. Female veterans have served within the AF for over 100 years. While their valuable contribution has been recognized, military culture, together with evolving Service requirements, have had a significant impact on the health and well-being of many. Yet, there is a dearth of evidence on the impact of alcohol use on female veteran health.

The limited existing evidence suggests that female veterans' alcohol use is increasing and that they are significantly more likely to report symptoms of hazardous drinking when compared with female civilians. Increased rates of hazardous drinking were also observed by Palmer and colleagues (202), who found that half (49%; n=389 of 779 female veterans) were misusing alcohol at a hazardous or higher level which is considered harmful to their health. To place this into context, the UK Chief Medical Officer recommends that everyone does not regularly drink more than 14 units per week, to keep health risks from drinking alcohol to a low level.

Alcohol misuse often co-occurs with common mental health disorders including PTSD, anxiety, or depression, and alcohol is frequently used as a coping mechanism. Common mental health disorders are more common in females than male veterans. Research has also shown that female veterans face barriers to accessing mental health support, often due to misusing alcohol. Ultimately, while female veterans drink less than male veterans, their rates of hazardous drinking are higher than the general population putting them at increased risk of poorer health.

The impact of alcohol misuse among female veterans on the wider society (e.g. health care utilization, productivity, and welfare) is unknown. In England, heavy drinking (deemed as drinking more than 14 units of alcohol per week) is estimated to cost the National Health Service (NHS) £3.5 billion per year (3.6% of its annual budget) and is more common in people with mental health difficulties, Since female veterans drink more than their civilian counterparts, the relative costs are likely to be even higher. Innovative solutions are urgently required.

In recent years there has been a growing treatment gap in the UK, with patients waiting longer for treatment and support for alcohol misuse. To overcome this gap, the investigators developed the DrinksRation platform (www.drinksration.app), an automated brief digital intervention designed to support help-seeking veterans in managing and reducing the amount they drink. DrinksRation is unique in that the app content is tailored using behaviour change techniques to promote positive changes in behaviour. DrinksRation is the only app targeting alcohol misuse in the UK AF. It is designed to (1) overcome geographical limitations; (2) use wearable technology (e.g. Fitbit, Apple Watch) to inform decision-making and personalization; (3) avoid the stigma associated with receiving help in person; and (4) provide convenience since users can use the app as they prefer (discretely or openly). The app is freely available via Apple and Google App stores. The app has received support and endorsement from Combat Stress and is currently being trialled in serving personnel. DrinksRation is supported by a robust evidence base, including a randomized controlled trial which demonstrated that the app is efficacious in reducing alcohol consumption.

The DrinksRation app was developed to support veterans who have sought help for a mental health problem and was not designed with potential gender differences in mind. A recent viewpoint highlighted a critical need for feminist intersectionality in digital health to incorporate the unique needs of females. Digital health technologies can bolster gender equality through increased access to healthcare, empowerment of one's health data, overcoming the specific barriers facing female veterans, and reducing the burden on healthcare systems.

This project aims to tailor the DrinksRation app to reflect the specific needs of female veterans and evaluate these changes using a confirmatory randomized controlled trial. It is hypothesized that a refined version of DrinksRation will be efficacious at reducing self-reported weekly alcohol consumption between baseline and 3-month follow-up (day 84) among female veterans who drink at a hazardous or harmful level.

ELIGIBILITY:
Inclusion criteria

* Are aged 18 years or older;
* Identify as female (self-reported sex);
* Live in the United Kingdom;
* Consume 15 UK units (approximately 150g) of alcohol or more per week as measured using Timeline Follow-back for alcohol consumption (TLFB; [23]) at baseline (day 0);
* Are veterans of the UK AF, defined as per UK definitions as having completed at least one day of paid employment in the UK AF (verified by self-report at eligibility screening);
* Have downloaded the mobile app onto an iOS or Android smartphone.

Exclusion criteria

-Does not own a smartphone phone.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Identify as female (self-reported sex);
Enrollment: 148 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Alcohol Use Change | 3 months
  The primary outcome measure is change between self-reported alcohol consumption as measured by the alcohol use 7-day timeline over the previous seven days between baseline (day 0) and 3-month follow-up (day 84). Outcome is reported as number of units, with a higher number of units indicating poorer outcome.

SECONDARY OUTCOMES:
Change in Alcohol use disorders identification test (AUDIT) | 3 months
  Changes in Alcohol Use Disorder Identification Test (AUDIT) score, measured at baseline (day 0) and day 84 follow-up between the control and intervention groups will be assessed. The AUDIT scale ranges from 0 to 40, with a higher scoring indicting poorer outcomes (ie. Higher scores means increased alcohol abuse).

CONTACTS AND LOCATIONS:
Locations (1):
- King's Centre for Military Health Research, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
All study data will be made available in an anonymized format alongside any source code via the Open Science Framework. There are no contractual agreements that limit access or sharing of data.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Upon publication of the main study report.
Access Criteria: None required.
URL: http://drinksration.app

REFERENCES:
- [Background] Leightley D, Rona RJ, Shearer J, Williamson C, Gunasinghe C, Simms A, Fear NT, Goodwin L, Murphy D. Evaluating the Efficacy of a Mobile App (Drinks:Ration) and Personalized Text and Push Messaging to Reduce Alcohol Consumption in a Veteran Population: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2020 Oct 2;9(10):e19720. doi: 10.2196/19720. PMID 33006569
- [Background] Williamson C, White K, Rona RJ, Simms A, Fear NT, Goodwin L, Murphy D, Leightley D. Smartphone-based alcohol interventions: A systematic review on the role of notifications in changing behaviors toward alcohol. Subst Abus. 2022;43(1):1231-1244. doi: 10.1080/08897077.2022.2074595. PMID 35670777
- [Background] Puddephatt JA, Leightley D, Palmer L, Jones N, Mahmoodi T, Drummond C, Rona RJ, Fear NT, Field M, Goodwin L. A Qualitative Evaluation of the Acceptability of a Tailored Smartphone Alcohol Intervention for a Military Population: Information About Drinking for Ex-Serving Personnel (InDEx) App. JMIR Mhealth Uhealth. 2019 May 24;7(5):e12267. doi: 10.2196/12267. PMID 31127726
- [Background] Leightley D, Puddephatt JA, Jones N, Mahmoodi T, Chui Z, Field M, Drummond C, Rona RJ, Fear NT, Goodwin L. A Smartphone App and Personalized Text Messaging Framework (InDEx) to Monitor and Reduce Alcohol Use in Ex-Serving Personnel: Development and Feasibility Study. JMIR Mhealth Uhealth. 2018 Sep 11;6(9):e10074. doi: 10.2196/10074. PMID 30206054
- [Background] Leightley D, Williamson C, Rona RJ, Carr E, Shearer J, Davis JP, Simms A, Fear NT, Goodwin L, Murphy D. Evaluating the Efficacy of the Drinks:Ration Mobile App to Reduce Alcohol Consumption in a Help-Seeking Military Veteran Population: Randomized Controlled Trial. JMIR Mhealth Uhealth. 2022 Jun 20;10(6):e38991. doi: 10.2196/38991. PMID 35724966
- [Derived] Williamson G, Carr E, Fear NT, Dymond S, King K, Simms A, Goodwin L, Murphy D, Leightley D. Digital Therapeutic Intervention for Women in the UK Armed Forces Who Consume Alcohol at a Hazardous or Harmful Level: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2023 Dec 19;12:e51531. doi: 10.2196/51531. PMID 38113103
- See also: Related Info — http://www.drinksration.app